CLINICAL TRIAL: NCT03215849
Title: The Effect of Biventricular Pacing in Heart Failure With Preserved Left Ventricular Ejection Fraction: A Pilot Mechanistic Analysis
Brief Title: Pacing in Heart Failure With Preserved LVEF
Acronym: MAPPLE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Cardiff Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 203878
Record Dates: First submitted 2017-06-22; First posted 2017-07-12 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine Medical Therapy (Sham Comparator): Routine Medical Therapy
  Interventions: Device: CRT-pacemaker device set to Routine Medical Therapy
- Routine Medical Therapy + LVP (Experimental): Routine Medical Therapy + LVP
  Interventions: Device: CRT-pacemaker device set to Routine Medical Therapy + LVP
- Routine Medical Therapy + BiVP (Experimental): Routine Medical Therapy + BiVP
  Interventions: Device: CRT-pacemaker device set to Routine Medical Therapy + BiVP

INTERVENTIONS:
Device: CRT-pacemaker device set to Routine Medical Therapy — Medtronic Serena™ QUAD CRT-P MRI™ SureScan™ W4TR05 set to Routine Medical Therapy
  Arms: Routine Medical Therapy
Device: CRT-pacemaker device set to Routine Medical Therapy + LVP — Medtronic Serena™ QUAD CRT-P MRI™ SureScan™ W4TR05 set to Routine Medical Therapy + LVP
  Arms: Routine Medical Therapy + LVP
Device: CRT-pacemaker device set to Routine Medical Therapy + BiVP — Medtronic Serena™ QUAD CRT-P MRI™ SureScan™ W4TR05 set to Routine Medical Therapy + BiVP
  Arms: Routine Medical Therapy + BiVP

SUMMARY:
A random-order cross-over pilot trial of a CE marked device (pacemaker) outside its current intended purposes.

The study will comprise 10 patients. Recruitment of patients will take place from The University Hospital of Wales (Cardiff & Vale University Health Board [CVUHB]). All patients recruited will have septal flattening during exercise demonstrated using contrast stress (exercise) echocardiography.

All 10 patients will be implanted with a CRT-pacemaker device and will be tested on all three of the following settings on separate visits (with a gap of up to 5 days between visits) in random order:

Routine Medical Therapy Routine Medical Therapy + LVP Routine Medical Therapy + BiVP

ELIGIBILITY:
Inclusion Criteria:

1. Clinical features consistent with heart failure. All patients will have symptoms of moderate to severe heart failure with New York Heart Association (NHYA) classification III or IV symptoms (for at least 3 months).
2. LV Ejection Fraction less or equal to 50%, with no evidence of significant valvular disease, no hypertrophic or restrictive cardiomyopathy, and no evidence of pericardial constriction.
3. Additionally all patients will have demonstrated evidence of septal flattening during exercise using contrast echocardiography.
4. Adults (over 18 years)
5. Negative test for Covid during surgical pre-assessment, and adherence to prescribed self-isolation before implantation.
6. Two weeks or more following final dose of vaccination against coronavirus.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Enrolment in other clinical studies.
3. BMI more than 35
4. Objective evidence of significant lung disease on formal lung function testing
5. Previous (within three months) or scheduled coronary revascularisation or other cardiac surgery
6. Acute coronary syndrome (within the previous three months)
7. History of atrial fibrillation (AF)
8. Renal insufficiency requiring haemodialysis
9. Life expectancy less than 6 months
10. Prosthetic heart valves
11. Blood coagulation disorders
12. Immunocompromised patients (e.g. AIDS, patients on steroids, cytotoxic drugs, and radiation therapy)
13. Currently pregnant, or intending to conceive.
14. Recent positive Covid test (up to 14 days prior to pre-assessment).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in septal radius of curvature (corrected for LV area) between rest and peak exercise on stress echocardiography across the three pacing states. | 12 weeks

SECONDARY OUTCOMES:
Change in LV area between rest and exercise across the three pacing states | 12 weeks
Change in Systolic and Diastolic mechanical Dyssynchrony Assessment on echocardiography across the three pacing states | 12 weeks
Change in rest and exercise E/E' on echocardiography across the three pacing states | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Yousef, Principal Investigator — Cardiff and Vale University Health Board
Locations (1):
- University Hospital Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No